CLINICAL TRIAL: NCT04189731
Title: Non-interventional Study Evaluating the Management of Pain Using a Technique Developed and Commonly Used by the Center, in Patients Who Underwent Arthroscopic Surgery of the Shoulder in the Outpatient Setting.
Acronym: BSS-CHIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Collaborators: Clinique chénieux (Unknown)
Responsible Party: Sponsor
Other Study IDs: 87RI19_0031 (BSS-CHIR)
Record Dates: First submitted 2019-12-02; First posted 2019-12-06 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Shoulder Pain
Keywords: Shoulder surgery; pain; suprascapular block
MeSH Terms: conditions — Shoulder Pain; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- supra-scapular block: Patient will have a short ISB (between 2h and 4h) relayed by a supra-scapular block (SSB) long (72h) through the placement of a perineural catheter thus allowing a continuous diffusion of Naropein® by an elastomeric pump

SUMMARY:
Shoulder surgery is performed usually under interscalene block considered as a gold standard. This anesthesia is well suited for hospitalized patients but not for outpatients. The Orthopedic Surgery Department of Clinique Chénieux has been operating patients requiring arthroscopic shoulder surgery with a short interscalene block relayed by a long suprascapular block. The main objective is to evaluate the effectiveness of this method by measuring the average pain over 3 days after the operation.

DETAILED DESCRIPTION:
The surgery of the shoulder is usually performed under interscalene block (ISB), considered as a gold standard. This anesthesia is well suited for hospitalized patients but not for outpatients. Indeed, the ISB entails, in addition to a sensory block, a motor block often useless and important since it extends beyond the shoulder to the entire upper limb. It can also be a source of anxiety and cause the risk of compression in the limb operated because of the extended sensorimotor block. It is also responsible for a painful bounce almost constant with sometimes the very rapid installation of intense pain when the effect of the sensory block disappears. This pain can be difficult to relieve despite frequent use of opioids.

The Orthopedic and Traumatologic Surgery Department of the Clinique Chénieux has been operating patients requiring arthroscopic surgery of the shoulder according to the following technique. It involves the establishment of a short ISB (between 2h and 4h) relayed by a supra-scapular block (SSB) long (72h) through the placement of a perineural catheter thus allowing a continuous diffusion of Naropein® by an elastomeric pump. The same day or the day after the operation, the patients return to their home and are followed by nurses.

The objective of this technique is to better manage postoperative pain, thus allowing the management of patients in outpatient surgery. A prospective non-interventional study will make it possible, in a context of common practice, to obtain data on the management of pain in operated patients and then to consider a generalization of this practice to other centers.

ELIGIBILITY:
Inclusion Criteria:

* Men, women between 18 and 70 years
* Patient in need of acromioplasty or rotator cuff surgery (ruptured cuff or calcification of the cuff) or reinsertion of the glenoid bead (Bankart intervention)
* Patient with an American Society of Anesthesiologists score (ASA) of 1 or 2

Exclusion Criteria:

* Patient needing shoulder surgery for other indications and open surgery
* Patient with cognitive impairment or dementia symptoms
* Patient with a BMI ≥ 35 without systemic morbidity requiring hospitalization
* Contraindication to the drugs used in the study (hypersensitivity to ropivacaine or other amide-bonded local anesthetics)
* Pregnant or lactating patient
* Patient with severe hepatic impairment
* Class III antiarrhythmic patient

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient in need of acromioplasty or rotator cuff surgery (ruptured cuff or calcification of the cuff) or reinsertion of the glenoid bead (Bankart intervention)
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Average of pain | Day1
  Score of average pain at D1, D2 and D3 by a numeric pain scale (NPS) <4/10
Average of pain | Day2
  core of average pain at D2 by a numeric pain scale (NPS) <4/10
Average of pain | Day 3
  core of average pain at D3 by a numeric pain scale (NPS) <4/10

SECONDARY OUTCOMES:
Number of readmissions | Day 7
  Number of readmissions the first week after the operation
Number of painful peaks | Day 0
  Number of painful peaks on awakening and leaving the block on the day of the operation
Analgesics consummation | Day 1, Day 2, Day 3, Day 4 and Day 7
  Amount and types of analgesics consumed / consumed non-opioid during the operation and the first week after the operation
Score of Pain | Day 4, Day 7, Day 15 and Day 30
  Score of minimum, maximum, average pain the month before the operation and by a numeric pain scale (NPS). Scale from 0 to 10.
Satisfied patient rate | Day 30
  Satisfied patient rate determined by using a satisfaction questionnaire with 4 responses: very satisfied, somewhat satisfied, somewhat dissatisfied and very dissatisfied
Number of postoperative complications | Month 3
  Number of postoperative complications at 3 month
Cartilaginous Toxicology | Month 6 and Month 12
  Cartilaginous Toxicology at 6 months and 12 months determined by radiograph of the shoulder of face in 3 rotations

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Chénieux, Limoges, France